CLINICAL TRIAL: NCT06892691
Title: Pleuroscopy First Versus Thoracentesis First in Patients With Suspected Malignant Pleural Effusions
Acronym: PERFECT-MPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Udit Chaddha, Associate Professor of Medicine and Thoracic Surgery, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY-24-00999
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-03

CONDITIONS: Pleural Effusion; Cancer
MeSH Terms: conditions — Pleural Effusion; Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to undergo either pleuroscopy first or thoracentesis first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pleuroscopy first (Active Comparator): Participants will undergo pleuroscopy first
  Interventions: Procedure: Pleuroscopy first
- Thoracentesis first (Active Comparator): Participants will undergo thoracentesis first
  Interventions: Procedure: Thoracentesis first

INTERVENTIONS:
Procedure: Pleuroscopy first — Pleuroscopies are performed under moderate sedation with local anesthesia. Through a 1-cm incision a camera is introduced into the pleural space and the space is inspected after draining all fluid. Targeted biopsies under direct visualization are obtained using forceps. The aspirated fluid and biopsies obtained are sent to the cytology and pathology laboratories for analysis.
  Arms: Pleuroscopy first
Procedure: Thoracentesis first — Thoracenteses are performed under local anesthesia with the insertion of a 5-8Fr catheter into the pleural space. The aspirated fluid obtained is sent to the cytology laboratory for analysis.
  Arms: Thoracentesis first

SUMMARY:
This is a randomized control trial of patients with suspected malignant pleural effusions to compare whether patients who have a thoracentesis or pleuroscopy (pleural biopsy) obtain an adequate biopsy, achieve a diagnosis, and begin cancer-directed therapy faster.

DETAILED DESCRIPTION:
This is a randomized control trial of patients with suspected malignant pleural effusions comparing patients who undergo either pleuroscopy or thoracentesis as the first diagnostic test. Both procedures are considered standard of care for this diagnosis but it is unknown which one provides more adequate biopsy samples and achieves faster diagnosis and shorter time to oncologic treatment. Currently, most patients undergo thoracentesis first and, if this is inadequate for diagnosis, they then undergo pleuroscopy for further biopsy samples. This study seeks to assess whether patients who undergo pleuroscopy as the first test obtain adequate biopsy samples and a faster path to further oncologic care compared to patients who undergo thoracentesis first. Patients will be recruited and randomized in a 1:1 manner.

Ultrasound is routinely used prior to the procedure and a chest x-ray is done after the procedure. Any other imaging will be determined by clinic need only. No imaging will be done for research purposes. No additional samples will be collected other than what is necessary for diagnostic purposes. In patients who have a non-diagnostic thoracentesis, the participants will be referred for pleuroscopy as the next diagnostic step. In the rare case that pleuroscopy does not achieve adequate diagnosis, the next step would be a liquid biopsy (non-invasive serologic testing for oncologic markers.) The need for liquid biopsy in participants in this study will be determined on a case-by-case basis depending on the clinical concern for malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Referral for diagnostic pleural procedure.
* Age ≥ 18 years.
* Suspected malignant pleural effusion (Suggestive radiologic appearance (based on computed tomography or positron emission tomography) OR suspected cancer with associated effusion.)

Exclusion Criteria:

* Inability to provide informed consent.
* Needs emergent drainage.
* Pleural effusion is known to be malignant.
* Suspected transudative, infectious or inflammatory effusion etiology.
* Having prior inconclusive/non-diagnostic thoracentesis or pleuroscopy.
* Patient is deemed by the clinical team to be more appropriate for VATS biopsy.
* Terminally ill patients in whom a diagnosis will not change management, or who is unlikely to be a candidate for oncological treatment due to significant comorbidities.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-03-24 (Actual); Primary Completion 2026-09-17 (Estimated); Study Completion 2026-09-17 (Estimated)

PRIMARY OUTCOMES:
Proportion of biopsies adequate for definitive diagnosis | 6 months
  Proportion of biopsies adequate for definitive diagnosis

SECONDARY OUTCOMES:
Time from initial visit with pulmonologist to procedure | 6 months
  Time from initial visit with pulmonologist to procedure
Time from initial procedure to diagnosis | 6 months
  Time from initial procedure to diagnosis
Time from initial visit with pulmonologist to diagnosis | 6 months
  Time from initial visit with pulmonologist to diagnosis
Time from initial visit with pulmonologist to seeing oncologist | 6 months
  Time from initial visit with pulmonologist to seeing oncologist
Time from initial visit with pulmonologist to starting treatment | 6 months
  Time from initial visit with pulmonologist to starting treatment
Time from seeing oncologist to starting treatment | 6 months
  Time from seeing oncologist to starting treatment
Frequency of procedure-related complications | 6 months
  Frequency of procedure-related complications
Frequency of additional diagnostic testing | 6 months
  Frequency of additional diagnostic testing

CONTACTS AND LOCATIONS:
Overall Officials: Udit Chaddha, MBBS, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (2):
- United States (2):
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  Any purpose. Proposals should be directed to udit.chaddha@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link tbd).